CLINICAL TRIAL: NCT04390243
Title: BrafPanc: A Phase II Trial of Binimetinib in Combination With Encorafenib in Patients With Pancreatic Malignancies and a Somatic BRAFV600E Mutation
Brief Title: Binimetinib and Encorafenib for the Treatment of Pancreatic Cancer in Patients With a Somatic BRAF V600E Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GI-1907; NCI-2020-02972 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI- 1907 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced Pancreatic Carcinoma; Metastatic Pancreatic Carcinoma; Recurrent Pancreatic Carcinoma; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — binimetinib; encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (encorafenib, binimetinib) (Experimental): Patients receive encorafenib PO QD and binimetinib PO BID on days 1-25. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Drug: Encorafenib

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162; Mektovi
Drug: Encorafenib — Given PO
  Other Names: Braftovi; LGX 818; LGX-818; LGX818

SUMMARY:
This phase II trial studies the side effects and how well the combination of binimetinib and encorafenib work in treating patients with pancreatic cancer with a somatic BRAF V600E mutation. Binimetinib and encorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving binimetinib and encorafenib may work better compared to the usual treatment in treating patients with pancreatic cancer and a somatic BRAF V600E mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of the combination of binimetinib and encorafenib as >= 2nd line of treatment for patients with metastatic pancreatic cancer with BRAF V600E mutation.

SECONDARY OBJECTIVES:

I. To determine in patients treated with the combination of binimetinib and encorafenib as >= 2nd line of treatment for patients with metastatic pancreatic cancer with BRAF V600E mutation:

Ia. The median progression-free survival. Ib. The median overall survival. Ic. Duration of response. Id. Time to response. Ie. The safety and tolerability.

OUTLINE:

Patients receive encorafenib orally (PO) once daily (QD) and binimetinib PO twice daily (BID) on days 1-25. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION:
* Histological confirmation of a pancreatic malignancy as confirmed by the local pathology lab
* Patients whose disease has progressed on (or who were intolerant of) at least one line of therapy for metastatic disease
* Patients whose disease has recurred with metastatic disease =< 12 weeks of completion of neoadjuvant or adjuvant systemic chemotherapy; or patients with locally advanced disease whose disease progressed to metastatic disease on, or =< 12 weeks after completion of systemic chemotherapy would also be eligible
* Provide informed written consent =< 28 days prior to pre-registration
* Central electronic/paper confirmation of the presence of a BRAF V600E mutation. This review is mandatory prior to pre-registration to confirm eligibility. Results from a Clinical Laboratory Improvement Act (CLIA)/College of American Pathologists (CAP) certified testing lab (commercial or institutional) that confirm the presence of a BRAF V600E mutation in the patient's tumor must be submitted for central review
* REGISTRATION: NOTE: Registration must occur =< 30 days after pre-registration
* Confirmation of the presence of BRAF V600E mutation in the patient's tumor
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2. (Form is available on the Academic and Community Cancer Research United [ACCRU] web site)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 14 days prior to registration)
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST) =< 2.5 x ULN; in participants with liver metastases =< 5 x ULN (obtained =< 14 days prior to registration)
* Aminotransferase (ALT) =< 2.5 x ULN; in participants with liver metastases =< 5 x ULN (obtained =< 14 days prior to registration)
* Calculated creatinine clearance must be >= 45 ml/min using the Cockcroft Gault formula (obtained =< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study). Note: During the active monitoring phase of a study (i.e., active treatment), participants must be willing to return to the consenting institution for follow-up
* Ability to swallow the investigational product tablets and capsules
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* REGISTRATION:
* Patients whose tumor harbors a BRAF non-V600E mutation or a BRAF fusion
* Prior therapy with BRAF inhibitor (e.g., encorafenib, dabrafenib, vemurafenib) and/or a MEK inhibitor (e.g., binimetinib, trametinib, cobimetinib)
* Known hypersensitivity or contraindication to any component of binimetinib or encorafenib or their excipients
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
  * NOTE: Female participants of childbearing potential must agree to use methods of contraception that are highly effective or acceptable, and to not donate ova from screening until 30 days after the last dose of study drug
  * NOTE: Male participants must agree to use methods of contraception that are highly effective or acceptable, and to not donate sperm from screening until 90 days after the last dose of study drug
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy. NOTE: Patients known to be human immunodeficiency virus ( HIV) positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 6 months prior to registration
* Left ventricular ejection fraction (LVEF) =< 50% as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO)
* Uncontrolled hypertension defined as persistent systolic blood pressure >= 150/100 mmHg or diastolic blood pressure >= 100 mmHg despite current therapy
* Triplicate average baseline corrected QT (QTc) interval >= 480 ms
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Patients who have had another active malignancy within the past two years are ineligible EXCEPT FOR patients with cervical cancer in situ, in situ carcinoma of the bladder, non-melanoma carcinoma of the skin, or patients who have had therapy with curative intent for breast or prostate cancer, but remain on adjuvant hormonal therapy
* Received anticancer therapy including chemotherapy, immunotherapy, or antineoplastic biologic therapy (e.g., erlotinib, cetuximab, bevacizumab etc.), =<14 days (=< 28 days for an antibody-based therapy) prior to registration
* Patients who have undergone major surgery (e.g., in-patient procedures) =< 6 weeks prior to registration or who have not recovered from side effects of such procedure
* Patients who have had radiotherapy =< 14 days prior to registration or who have not recovered from side effects of such procedure. NOTE: Palliative radiation therapy must be complete 7 days prior to the first dose of study treatment
* Patient has not recovered to =< grade 1 from toxic effects of prior therapy before registration. EXCEPTIONS: Stable chronic conditions (=< grade 2) that are not expected to resolve (such as neuropathy, myalgia, alopecia, prior therapy-related endocrinopathies)
* Uncontrolled or symptomatic brain metastases or leptomeningeal carcinomatosis that are not stable, require steroids, are potentially life-threatening or have required radiation =< 28 days prior to registration.

  * NOTE: Patients with previously treated brain metastases may participate provided they are stable (e.g., without evidence of progression by radiographic imaging for =< 28 days prior to registration and neurologic symptoms have returned to baseline), and have no evidence of new or enlarging brain metastases or central nervous system (CNS) edema, and does not require steroids at least 7 days before the first dose of study treatment.
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of study drug (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal absorption), or recent (=< 12 weeks) history of a partial or complete bowel obstruction, or other condition that will interfere significantly with the absorption or oral drugs
* Known history of acute or chronic pancreatitis
* Concurrent neuromuscular disorder that is associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amytrophic lateral sclerosis, spinal muscular atrophy)
* History or current evidence of RVO or current risk factors for retinal vein occlusion (RVO) (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease
* Current use of prohibited medication (including herbal medications, supplements, or foods), or use of prohibited medication =< 7 days prior to registration
* History of thromboembolic or cerebrovascular events =< 12 weeks prior to registration. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli.

  * NOTE: Patients with either deep vein thrombosis or pulmonary emobli that do not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for =< 4 weeks prior to registration
  * NOTE: Patients with thromboembolic events related to indwelling catheters or other procedures may register
* Evidence of hepatitis B Virus (HBV) or hepatitis C Virus (HCV) infection.

  * NOTE: Patients with laboratory evidence of cleared HBV or HCV infection may register.
  * NOTE: Patients with no prior history of HBV infection who have been vaccinated against HBV and who have a positive antibody against hepatitis B surface antigen as the only evidence of prior exposure may register

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Hendifar, Principal Investigator — Academic and Community Cancer Research United
Locations (5):
- United States (5):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Encorafenib, Binimetinib): Patients receive encorafenib PO QD and binimetinib PO BID on days 1-25. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.> > Binimetinib: Given PO>
  > Encorafenib: Given PO
Period: Overall Study
Arm/Group | Treatment (Encorafenib, Binimetinib)
Started | 6
Completed | 0
Not Completed | 6
Not completed — Death | 1
Not completed — Disease Progression | 4
Not completed — Patient was on treatment when study was terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Encorafenib, Binimetinib)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Line of Treatment [Count of Participants; unit: Participants] — 2nd line - patients received study treatment as their 2nd line of therapy 3rd line - patients received study treatment as their 3rd line of therapy
  Participants
    2nd line | 4
    3rd line | 2
Histologic Grade of Malignancy [Count of Participants; unit: Participants] — * G1 (Well differentiated)
  * G2 (Moderately differentiated)
  * GX (Grade cannot be assessed)
  G1 is associated with better prognosis, G3 is associated with poorer prognosis
  Participants
    G1 | 1
    G2 | 3
    GX | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) at 24 Weeks
Description: An objective response is defined as a complete or partial response with a confirmation scan not less than 4 weeks after the initial scan. Disease status will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria. The final ORR point estimate and corresponding 95% confidence interval will be reported.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Treatment (Encorafenib, Binimetinib): Patients receive encorafenib PO QD and binimetinib PO BID on days 1-25. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.
  >
  > Binimetinib: Given PO
  >
  > Encorafenib: Given PO
Arm/Group | Treatment (Encorafenib, Binimetinib)
Number analyzed (Participants) | 6
percentage of patients | 33.33 [4.33 to 77.72]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from registration to clinical or radiographic disease progression or death, whichever occurs first, as defined by RECIST 1.1 criteria. PFS will be estimated using the Kaplan-Meier method. The median PFS and corresponding 95% confidence interval will be reported.
Time Frame: 25 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Encorafenib, Binimetinib)
Number analyzed (Participants) | 6
months | 7.1 [1.7 to NA] — The upper limit of the confidence interval was not estimatable due to an insufficient number of participants with events

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from registration to death from any cause. OS will be estimated using the Kaplan-Meier method. The median overall survival and corresponding 95% confidence interval will be reported.
Time Frame: 25 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Encorafenib, Binimetinib)
Number analyzed (Participants) | 6
months | 15.0 [3.1 to NA] — The upper limit of the confidence interval was not estimatable due to an insufficient number of participants with events

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the duration of time from first documentation of an objective response to the earliest date disease progression is documented or death from any cause. Duration of response will be estimated using the Kaplan-Meier method. The median duration of response and corresponding 95% confidence interval will be reported.
Time Frame: 12 months
Population: Only patients that achieved an objective response within 12 months were included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Encorafenib, Binimetinib)
Number analyzed (Participants) | 3
months | 9.9 [8.5 to NA] — The upper limit of the confidence interval was not estimatable due to an insufficient number of participants with events

5. Secondary Outcome: Time to Response
Description: Time to response is defined as the duration of time from registration to the first documentation of an objective response. Time to response will be estimated using the Kaplan-Meier method. The median time to response and corresponding 95% confidence interval will be reported.
Time Frame: 25 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Encorafenib, Binimetinib)
Number analyzed (Participants) | 6
months | 3.9 [3.6 to NA] — The upper limit of the confidence interval was not estimatable due to an insufficient number of participants with events

6. Secondary Outcome: Number of Patients With Grade 3+ Adverse Events
Description: Adverse Events as defined by National Institute of Health (NIH) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. All patients who have initiated treatment will be considered evaluable for adverse event analyses. The rate of patients experiencing a grade 3+ adverse event will be reported.
Time Frame: 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Encorafenib, Binimetinib)
Number analyzed (Participants) | 6
Participants | 3

ADVERSE EVENTS:
Time Frame: 25 months
Groups:
- Treatment (Encorafenib, Binimetinib): Patients receive encorafenib PO QD and binimetinib PO BID on days 1-25. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.
  * Binimetinib: Given PO
  * Encorafenib: Given PO
Arm/Group | Treatment (Encorafenib, Binimetinib)
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Encorafenib, Binimetinib) (N=6)
Disease progression (General disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Encorafenib, Binimetinib) (N=6)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 2 (14)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (44)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
CPK increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (8)
Weight gain (Investigations) | 1 (3)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (13)
Headache (Nervous system disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (3)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT04390243/Prot_SAP_000.pdf